CLINICAL TRIAL: NCT05535712
Title: Pilot Study of Single Port Robotic Surgery for Anatomical Lung Resection
Brief Title: Single Port Robotic Lung Anatomical Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202101423A0
Record Dates: First submitted 2022-06-07; First posted 2022-09-10 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Robotic Surgical Procedure
Keywords: Early Stage Lung Cancer; Da Vinci SP; Robotic Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: clinical lung cancer who receive Da Vinci sp robotic surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Da Vinci SP intervnetion group (Experimental): for patients who received Da Vinci SP robotic surgery
  Interventions: Device: Lung Anatomic Resection (Da Vinci SP)

INTERVENTIONS:
Device: Lung Anatomic Resection (Da Vinci SP) — To evaluate the performance and safety of the da Vinci SP® Surgical System in anatomical lung resection

SUMMARY:
This is the first human clinical study for explore the feasibility of lung anatomic resection through Da Vinci SP surgical platform

DETAILED DESCRIPTION:
During the past several years, minimally invasive thoracic surgery has evolved from thoracoscopic approaches using 3 -4 ports to a single incision video-assisted thoracoscopic surgery (VATS) techniques. Recently, the experience acquired with the uniportal VATS technique through the intercostal space has allowed the development of a uniportal VATS subxiphoid or subcostal approach for major pulmonary resections. The advantage of using a subxiphoid or subcostal entry is to reduce pain by avoiding possible trauma of intercostal nerves caused by thoracic incisions. However, the longer distance from the subxiphoid or subcostal incision to the hilum makes this approach more difficult to perform anatomical pulmonary resections.During this same period of evolution into uniportal VATS surgery, robotic thoracic surgery has gained popularity as an alternative to traditional VATS. The advantages of robotics are the ability to perform surgery more precisely with articulated or wristed instruments, motion scaling, and tremor filtration, as well as improved visualization thanks to 3D high-definition video. However, currently 4 -5 incisions are still necessary to perform anatomic robotic resections.Recently, there has been a convergence of these two trends-uniportal surgery and robotic-assisted surgery-and has resulted in a single port robotic system, the da Vinci SP by Intuitive Surgical Cooperation. For this new platform, investigators plan to practice in thoracic anatomic lung resection

ELIGIBILITY:
Inclusion Criteria:

1. Age >20 and <75 years-old
2. Willing and able to provide informed consent
3. ASA≤ 3
4. The subject is undergoing the following procedures

   1. diagnosis with of clinical stage I lung cancer
   2. The primary tumor should be less than ≤4cm diameter and ≥ 2 cm away from the origin of the associated lobar bronchus
5. Preoperative platelet count 150-400 (1000/ uL)

Exclusion Criteria:

1. Congestive heart failure (NHYA > II)
2. Subjects with a known bleeding or clotting disorder
3. Subjects actively receiving therapeutic dose anticoagulation or anti-platelet medications at the time of operation
4. Subjects under immunomodulatory or immunosuppressive regimen (e.g. transplant patient, steroid requirement) within 30 days prior to the planned surgery
5. Subjects with pulmonary hypertension
6. In need of extended resection (e.g. Chest wall, Carina, major vessel, bilobectomy) and reconstruction (e.g. Sleeve resection, bronchoplasty, angioplasty)
7. Previous ipsilateral thoracic surgery or sternotomy
8. Uncontrolled illness 6 months prior to planned surgical procedure including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
9. Previous neoadjuvant medical and/or radiation therapy
10. Subject has a contraindication for general anesthesia or surgery
11. Life expectancy < 6 months
12. Anatomy determined intra-operatively to be unsuitable for minimally invasive surgery
13. Subjects belong to vulnerable population (e.g., pregnancy or breastfeeding)
14. International normalized ratio, INR >1.4
15. Activated Partial Thromboplastin Time , APTT >35 -

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of conversion rate | During Surgery
  The primary performance endpoint will be assessed as the ability to successfully complete the planned anatomic resection procedure with the da Vinci SP System, with no conversion to thoracoscopic, multi-port robotic, or open surgery. Usage of additional assistant port(s) is not considered a conversion.

SECONDARY OUTCOMES:
Incidence of Treatment Related Adverse Events | One Year
  The primary safety endpoint will be assessed as the incidence of all intra-operative and post-operative adverse events that occur within the study follow-up period. Complications are assessed using the Common Terminology Criteria for Adverse Events, CTCAE.
Peri-operative parameters | From Surgery to ward,2- day
  Operation time (minute), docking time (minute), console time(minute), anesthesia time(minute), Time from recovery room to ward (minute)
Peri-operative parameters: blood loss related | During surgery
  which include bloods loss(ml) during operation, blood transfusion (ml) during surgery
Hospitalization parameters | During Hospitalization, an average of 4 days
  which include, length of hospital stay (day)
Operative related complications during hospitalization | During Hospitalization, an average of 4 days
  which include in-hospital mortality and morbidity, reasons need for reoperation, unplanned procedure after surgery
Patient disposition immediately after surgery | During Hospitalization, an average of 1 day
  ICU, ward

OTHER OUTCOMES:
30-day follow-up | Post-operative data through 30-day follow-up
  Complications (assed according to CTCAE)
Questionnaire assessment (1) | Through study completion, an average of 1 year
  Enrolled subjects would be assessed by pain scale score at baseline (preoperatively), during inpatient phase.
  Neuropathic pain assessment (Assessment of post-VATS surgery neuralgia- pain DETECT Questionnaire), performed during inpatient phase (Post-operation 1 day, 2 days and day of discharge) and 1 week, 1,3,6,12 months after discharge.
Questionnaire assessment (2) | Through study completion, an average of 1 year
  Enrolled subjects would be assessed by numbness score at baseline (preoperatively), during inpatient phase.
  Neuropathic pain assessment (Assessment of post-VATS surgery neuralgia- pain DETECT Questionnaire), performed during inpatient phase (Post-operation 1 day, 2 days and day of discharge) and 1 week, 1,3,6,12 months after discharge.
90-day follow up (1) | Post-operative data through 90-day follow-up
  Complications (assed according to CTCAE)
Pathological Report | Post-operative data through 30-day follow-up
  pathologic tumor staging, surgical margins
90-day Follow up (2) | Post-operative data through 90-day follow-up
  Unplanned procedure-related reoperations or readmissions, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Yin Kai Chao, MD,PHD, Principal Investigator — CHENG GUNG MEMORIAL HOSPITAL
Locations (1):
- Chang Gung Memeorial Hospital, Linkou Medical Center, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng C, Tagkalos E, Ng CB, Hsu YC, Huang YY, Wu CF, Chao YK. Subcostal uniportal robotic anatomic lung resection: A pilot trial. JTCVS Tech. 2024 Apr 28;25:160-169. doi: 10.1016/j.xjtc.2024.01.024. eCollection 2024 Jun. PMID 38899114